CLINICAL TRIAL: NCT03471260
Title: Phase Ib/II Investigator Initiated Study of the IDH1-Mutant Inhibitor Ivosidenib (AG120) With the BCL2 Inhibitor Venetoclax +/- Azacitidine in IDH1-Mutated Hematologic Malignancies
Brief Title: Ivosidenib and Venetoclax With or Without Azacitidine in Treating Patients With IDH1 Mutated Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0490; NCI-2018-00921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0490 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-03-02; First posted 2018-03-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Hematopoietic and Lymphoid System Neoplasm; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Azacitidine; ivosidenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, ivosidenib, azacitidine) (Experimental): Patients receive venetoclax PO daily on days 1-14. Patients also receive ivosidenib PO daily on days 15-28 of cycle 1 and days 1-28 of subsequent cycles. Patients may also receive azacitidine IV over 30-60 minutes or SC on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Ivosidenib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of venetoclax and how well it works when given together with ivosidenib with or without azacitidine, in treating patients with IDH1-mutated hematologic malignancies. Venetoclax and ivosidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ivosidenib and venetoclax with azacitidine may work better in treating patients with hematologic malignancies compared to ivosidenib and venetoclax alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability, maximum tolerated dose (MTD), and recommended phase 2 dose (RP2D) of the combination of ivosidenib with venetoclax, with or without the addition of azacitidine, in IDH1-mutated patients with advanced hematologic malignancies. (Phase Ib) II. To determine the overall response rate (ORR) including complete response (CR), CR with incomplete blood count recovery (CRi), morphologic leukemia-free state (MLFS), and partial response (PR) of the combination of ivosidenib and venetoclax, with or without the addition of azacitidine, in IDH1-mutated patients with acute myeloid leukemia (AML). (Phase II)

SECONDARY OBJECTIVES:

I. Characterize the pharmacokinetic (PK) profiles of venetoclax and ivosidenib in combination in plasma samples (in Part 1b).

II. To evaluate molecular and cellular biomarkers that may be predictive of antitumor activity and/or resistance to treatment including evaluation of 2HG, IDH1 VAF levels before, during and after treatment.

III. To determine time to event endpoints including duration of response (DOR), event free survival (EFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Evaluate minimal residual disease (MRD) using multiparameter flow cytometry, cytogenetics and molecular evaluation.

II. Evaluate global gene expression profiles, deoxyribonucleic acid (DNA) methylation profiles, BH3 profiling and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

OUTLINE: This is a phase Ib, dose-escalation study of venetoclax followed by a phase II study.

Patients receive venetoclax orally (PO) daily on days 1-14. Patients also receive ivosidenib PO daily on days 15-28 of cycle 1 and days 1-28 of subsequent cycles. Patients may also receive azacitidine intravenously (IV) over 30-60 minutes or subcutaneously (SC) on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then monthly for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. ECOG performance status of < 2.
3. IDH1-R132 mutated disease status as assessed by local laboratory. 2HG-producing IDH1 variants outside of R132 (i.e. R100) may be eligible after discussion with the PI.
4. Relapsed/refractory AML, or treatment-naïve patients with AML who are not eligible for standard induction chemotherapy. Patients with high-risk MDS, MDS/MPN or MPN (defined as > 10% bone marrow blasts, or intermediate or high risk by IPSS, R-IPSS or D-IPSS) that have failed standard therapy may also be eligible after discussion with the PI.
5. Adequate hepatic function (direct bilirubin < 2 x ULN, ALT and/or AST < 3x ULN) unless deemed to be related to underlying leukemia.
6. Adequate renal function including creatinine clearance > 30 ml/min based on the Cockcroft-Gault equation.
7. Willing and able to provide informed consent
8. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 7 days for cytotoxic or non-cytotoxic (immunotherapy) agents.
9. Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug.

Exclusion Criteria:

1. Patients with known allergy or hypersensitivity to ivosidenib or venetoclax.
2. Patients who have previously received either ivosidenib or venetoclax.
3. Patients with any concurrent uncontrolled clinically significant medical condition including infection, laboratory abnormality, or psychiatric illness, which could place the patient at unacceptable risk of study treatment.
4. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea and/or one dose of cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy.
5. Patients receiving concomitant strong CYP3A inducers (avasimibe, carbamazepine, phenytoin, rifampin, rifabutin, St. John's wort) within 3 days of start of study therapy.
6. Patients with active graft-versus-host-disease (GVHD) status post stem cell transplant (patients without active GVHD on chronic suppressive immunosuppression and/or phototherapy for chronic skin GVHD are permitted after discussion with the PI).
7. Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
8. Patients with a concurrent active malignancy under treatment.
9. QTc interval using Fridericia's formula (QTcF) > 450 msec. Bundle branch block and prolonged QTc interval are permitted after discussion with the PI.
10. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known HIV infection.
11. Subject has a white blood cell count > 25 x 10⁹/L. (Note: Hydroxyurea is permitted to meet this criterion.)
12. Nursing women, women of childbearing potential (WOCBP) with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception a. Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, IUD, and double barrier methods (for example a condom in combination with a spermicide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  Defined as complete response (CR), CR with incomplete blood count recovery (CRi), morphologic leukemia-free state (MLFS), and partial response (PR) based on revised International Working Group (IWG) response criteria. Analysis will be performed for enrolled subjects.
Incidence of adverse events | Up to 3 years
  Will be collected using leukemia adverse event guidelines.
Dose-limiting toxicity | Up to 56 days
  Defined as any grade 3 or 4, clinically significant non-hematologic adverse event or abnormal laboratory value.

SECONDARY OUTCOMES:
Response to therapy | Up to 3 years
  Will be calculated.
Duration of response | From the date of initial response to first documented disease progression/relapse or death, assessed up to 3 years
  Will be calculated.
Event-free survival | From treatment initiation to date of documented treatment failure, relapse, or death from any cause, assessed up to 3 years
  Will be calculated.
Overall survival | Up to 3 years
  Will be calculated.

OTHER OUTCOMES:
Plasma concentrations and pharmacokinetic parameter | Up to 3 years
  Will be tabulated for each subject, visit, and dose level, and summary statistics will be computed for each sampling time and each parameter.
Peripheral blood and bone marrow aspirate samples | Up to 3 years
  Biomarker assays may include, but are not limited to, BH3 profiling and characterization of BCL-2 and related proteins, IDH1 mutant status, serum R-2HG analysis, and assessment of the depth of response and monitoring of disease recurrence by assessment of minimal residual disease in the bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] DiNardo CD, Marvin-Peek J, Loghavi S, Takahashi K, Issa GC, Jen WY, Daver NG, Reville PK, Short NJ, Sasaki K, Mullin JK, Bradley CA, Borthakur G, Maiti A, Alvarado Y, Pemmaraju N, Abbas HA, Hammond DE, Haddad F, Bravo GM, Chien KS, Yilmaz M, Kornblau SM, Jabbour E, Ravandi F, Kadia T, Garcia-Manero G, Konopleva MY, Kantarjian HM. Outcomes of Frontline Triplet Regimens With a Hypomethylating Agent, Venetoclax, and Isocitrate Dehydrogenase Inhibitor for Intensive Chemotherapy-Ineligible Patients With Isocitrate Dehydrogenase-Mutated AML. J Clin Oncol. 2025 Aug 20;43(24):2692-2699. doi: 10.1200/JCO-25-00640. Epub 2025 Jun 13. PMID 40513054
- [Derived] Wilde L, Kasner M. Whom should we treat with novel agents? Specific indications for specific and challenging populations. Hematology Am Soc Hematol Educ Program. 2021 Dec 10;2021(1):24-29. doi: 10.1182/hematology.2021000228. PMID 34889407
- See also: M D Anderson Cancer Center — http://www.mdanderson.org